CLINICAL TRIAL: NCT00000979
Title: Comparison of 2',3'-Dideoxyinosine (ddI) (BMY-40900) and Zidovudine in Therapy of Patients With HIV Infection
Brief Title: Comparison of ddI Versus Zidovudine in HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry)
Purpose: Treatment
Other Study IDs: ACTG 116; 070V1; ACTG 116-A; ACTG 116-B/117; AI454-008
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2003-01

CONDITIONS: HIV Infections
Keywords: Didanosine; Zidovudine
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine; Didanosine

INTERVENTIONS:
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To compare the effectiveness and toxicity of didanosine (ddI) and zidovudine (AZT) in patients with AIDS, advanced AIDS-related complex (ARC), or asymptomatic infection with CD4 counts < 200 cells/mm3.

AZT is effective in reducing mortality in patients with AIDS who receive the drug after the first episode of Pneumocystis carinii pneumonia (PCP) and in patients with advanced ARC. However, AZT therapy has been associated with significant toxicities. In addition, the effectiveness of AZT appears to decrease during the second and third years of therapy. For these reasons, the development of alternative therapy that would be at least as effective but less toxic is of great importance. The drug ddI is an antiviral agent that inhibits replication (reproduction) of HIV with less apparent toxicity than AZT.

DETAILED DESCRIPTION:
AZT is effective in reducing mortality in patients with AIDS who receive the drug after the first episode of Pneumocystis carinii pneumonia (PCP) and in patients with advanced ARC. However, AZT therapy has been associated with significant toxicities. In addition, the effectiveness of AZT appears to decrease during the second and third years of therapy. For these reasons, the development of alternative therapy that would be at least as effective but less toxic is of great importance. The drug ddI is an antiviral agent that inhibits replication (reproduction) of HIV with less apparent toxicity than AZT.

AMENDED: 9/28/90 Patients are assigned to one of 2 treatments under a double-blind, randomly allocated, experimental design if their duration of prior AZT therapy is 0 to 16 weeks. (Patients who entered with no more than 16 weeks prior AZT and who were randomized to ddI will continue to be dosed at that level, adjusted for weight, and followed as originally planned.) Patients are assigned to one of 3 treatments as explained prior to this amendment if their duration of prior to AZT therapy is greater than 16 weeks. Original design: Patients are assigned to one of three treatments under a double-blind randomly allocated experimental design. ddI will be administered at two dose levels.

It is anticipated that patients will be seen as outpatients every 2 weeks for the first 4 weeks of the study and monthly thereafter. This study continues for at least 18 months after the entry of the first subject.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* Aerosolized pentamidine (300 mg every 4 weeks using a Respirgard II nebulizer). In the event of physiological intolerance, alternative prophylaxis may be: Trimethoprim / sulfamethoxazole 1 DS tab per day or dapsone 50 - 100 mg/day.

Allowed:

Maintenance therapy for active AIDS defining opportunistic infections for patients with 9 to 47 weeks' experience with zidovudine (AZT).

Treatment of opportunistic infections with other than sulfonamide containing drugs:

* Pyrimethamine and sulfadiazine or clindamycin for suppression of toxoplasmosis acquired after study entry; fluconazole or amphotericin B for suppression of cryptococcosis or ketoconazole for candidiasis.

Intravenous acyclovir for up to 10 days. Erythropoietin for patients under the relevant treatment IND. Analgesics, antihistamines, antiemetics, antidiarrheal agents for symptomatic therapy for toxicities.

Isoniazid (INH) if no other acceptable therapy is available.

Metronidazole may be used for single courses of therapy not to exceed 14 days within consecutive 90 day intervals. Note:

* Ketoconazole and dapsone should be taken 2 hours before or 2 hours after taking ddI (amendment 5/20/91).

Concurrent Treatment:

Allowed:

* Blood transfusions for hemoglobin toxicity.

Patients must:

* Have a diagnosis of AIDS or advanced AIDS related complex (ARC), or per 8/09/90 amendment, asymptomatic HIV infection with CD4 count = or < 200 cells/mm3.
* Be either naive to zidovudine (AZT) or have taken AZT for = or < 48 weeks.
* Have ended treatment for acute Pneumocystis carinii pneumonia (PCP) at least 2 weeks before study entry. For patients with 2 months or less experience with AZT, PCP infection will be the single and only AIDS-defining infection and must have been within 120 days of study entry. Per amendment, other AIDS-defining conditions are allowed in the 8 weeks prior to study entry (for patients in the AZT stratum).Only one episode of PCP is permitted unless patient has > 2 months AZT experience in which case > 1 prior episode of PCP infection is allowed.
* Not have experienced a major intolerance to AZT at doses of at least 500 mg if the patient was on AZT therapy for = or < 48 weeks. A major intolerance is defined as recurrent grade 3 or greater toxicity which results in discontinuation of drug.

Allowed:

* Basal cell carcinoma.
* In situ carcinoma of the cervix.
* Occasional premature atrial or ventricular contraction.
* Patients developing new opportunistic infections after study entry will remain on this protocol.
* Patients whose AIDS-defining condition is Kaposi's sarcoma alone must have CD4 cell counts < 300 cells/mm3.

Prior Medication:

Allowed:

* Previous treatment with zidovudine (AZT) up to 48 weeks.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or diseases are excluded:

* Kaposi's sarcoma (KS) with evidence of visceral disease or where KS requires chemotherapy; subjects with localized KS having CD4 counts = or > 200 cells/mm3.
* AIDS-dementia complex = or > stage 2.
* Prior history of acute pancreatitis within past 2 years or chronic pancreatitis.
* Intractable diarrhea.
* History of seizures within past 6 months or currently requiring anticonvulsants for control.
* History of past or current heart disease.
* Presence of a malignancy likely in the investigators opinion to require cytotoxic myelosuppressive chemotherapy during the expected course of this trial.

Concurrent Medication:

Excluded:

* Oral acidifying agents.
* Neurotoxic drugs. NOTE: If patients require therapy for PCP with IV pentamidine, study mediation is stopped.

Patients with the following are excluded:

* Active AIDS defining events. Maintenance therapy for prior AIDS-defining opportunistic infections is permitted.
* Intolerance to AZT at doses of 500 mg because of recurrent grade 3 toxicity or greater which resulted in discontinuation of drug.
* Neoplasms not specifically allowed.
* Previous enrollment in any study of ddI, ddC or d4T.
* > 48 weeks of AZT therapy.
* An opportunistic infection not adequately controlled with suppressive therapies allowed in the protocol.
* Psychological or emotional problems sufficient, in the investigator's opinion, to prevent adequate compliance study therapy.
* Life expectancy = or < 6 months.

Prior Medication:

Excluded:

* Ganciclovir.
* AZT for = or > 48 weeks.

Excluded within 14 days of study entry:

* Erythropoietin (Eprex).

Excluded within 30 days of study entry:

* Anti-HIV therapy other than AZT.
* Biologic response modifiers.
* Other investigational drugs.
* Corticosteroids.
* Neurotoxic drugs.

Excluded within 90 days of study entry:

* Ribavirin.

Prior Treatment:

Excluded within 14 days of study entry:

* Transfusion.

Active alcohol or drug abuse sufficient, in the investigator's opinion, to prevent adequate compliance with study therapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500
Dates: Primary Completion 1992-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R Dolin, Study Chair; M Fischl, Study Chair
Locations (71):
- United States (70):
  - Children's Hosp of Los Angeles/UCLA Med Ctr, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Palo Alto Veterans Adm Med Ctr / Stanford Univ, Palo Alto, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Stanford Univ School of Medicine, Stanford, California
  - Olive View Med Ctr, Sylmar, California
  - Sepulveda Veterans Adm Med Ctr / Olive View Med Ctr, Sylmar, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Mountain States Regional Hemophilia Ctr / Univ of Colorado, Denver, Colorado
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Whitman - Walker Clinic, Washington D.C., District of Columbia
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - G E Morey Jr, Fort Lauderdale, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Edward Hines Veterans Administration Hosp, Hines, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Louisiana Comprehensive Hemophilia Care Ctr, New Orleans, Louisiana
  - Louisiana State Univ Med Ctr / Tulane Med School, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Med Ctr of Central Massachusetts, Worcester, Massachusetts
  - Univ of Massachusetts Med Ctr, Worcester, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - Nebraska Regional Hemophilia Ctr, Omaha, Nebraska
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - City Hosp Ctr at Elmhurst / Mount Sinai Hosp, Elmhurst, New York
  - Beth Israel Med Ctr / Peter Krueger Clinic, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - SUNY - Stony Brook, Stony Brook, New York
  - SUNY / State Univ of New York, Syracuse, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Bronx Veterans Administration / Mount Sinai Hosp, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Bowman Gray School of Medicine / Wake Forest Univ, Winston-Salem, North Carolina
  - Holmes Hosp / Univ of Cincinnati Med Ctr, Cincinnati, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Med College of Ohio, Toledo, Ohio
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Hemophilia Ctr of Western PA / Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Univ of Pittsburgh Med School, Pittsburgh, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Tennessee / E Tennessee Comprehensive Hemophilia Ctr, Knoxville, Tennessee
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Hermann Hosp / Univ Texas Health Science Ctr, Houston, Texas
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
  - Univ of Utah School of Medicine, Salt Lake City, Utah
  - Dr Stephen L Green, Hampton, Virginia
  - Univ of Washington, Seattle, Washington
  - Dr Brian Buggy, Milwaukee, Wisconsin
  - Milwaukee County Med Complex, Milwaukee, Wisconsin
  - Great Lakes Hemophilia Foundation, Milwaukee, Wisconsin
- San Juan Veterans Administration Med Ctr, San Juan, Puerto Rico

REFERENCES:
- [Background] Dolin R, Amato DA, Fischl MA, Pettinelli C, Beltangady M, Liou SH, Brown MJ, Cross AP, Hirsch MS, Hardy WD, et al. Zidovudine compared with didanosine in patients with advanced HIV type 1 infection and little or no previous experience with zidovudine. AIDS Clinical Trials Group. Arch Intern Med. 1995 May 8;155(9):961-74. PMID 7726705
- [Background] Bozzette SA, Hays RD, Berry SH, Kanouse DE. A Perceived Health Index for use in persons with advanced HIV disease: derivation, reliability, and validity. Med Care. 1994 Jul;32(7):716-31. doi: 10.1097/00005650-199407000-00005. PMID 8028406
- [Background] Fiscus SA, Heggem-Snow A, Troiani L, Wallmark E, Folds JD, Sheff B, van der Horst CM. Transient high titers of HIV-1 in plasma and progression of disease. J Acquir Immune Defic Syndr Hum Retrovirol. 1995 May 1;9(1):51-7. PMID 7712235
- [Background] Schooley RT. Correlation between viral load measurements and outcome in clinical trials of antiviral drugs. AIDS. 1995 Dec;9 Suppl 2:S15-S19. PMID 8775802
- [Background] Kozal MJ, Kroodsma K, Winters MA, Shafer RW, Efron B, Katzenstein DA, Merigan TC. Didanosine resistance in HIV-infected patients switched from zidovudine to didanosine monotherapy. Ann Intern Med. 1994 Aug 15;121(4):263-8. doi: 10.7326/0003-4819-121-4-199408150-00005. PMID 7518658
- [Background] Fichtenbaum CJ, Clifford DB, Powderly WG. Risk factors for dideoxynucleoside-induced toxic neuropathy in patients with the human immunodeficiency virus infection. J Acquir Immune Defic Syndr Hum Retrovirol. 1995 Oct 1;10(2):169-74. doi: 10.1097/00042560-199510020-00009. PMID 7552481
- [Background] Spino C, Kahn JO, Dolin R, Phair JP. Predictors of survival in HIV-infected persons with 50 or fewer CD4 cells/mm3. J Acquir Immune Defic Syndr Hum Retrovirol. 1997 Aug 15;15(5):346-55. doi: 10.1097/00042560-199708150-00004. PMID 9342254
- [Result] Richardson D, Liou SH, Kahn JO. Uric acid and didanosine compliance in AIDS clinical trials: an analysis of AIDS Clinical Trials Group protocols 116A and 116B/117. J Acquir Immune Defic Syndr (1988). 1993 Nov;6(11):1212-23. PMID 8229656
- [Result] Welles SL, Jackson JB, Yen-Lieberman B, Demeter L, Japour AJ, Smeaton LM, Johnson VA, Kuritzkes DR, D'Aquila RT, Reichelderfer PA, Richman DD, Reichman R, Fischl M, Dolin R, Coombs RW, Kahn JO, McLaren C, Todd J, Kwok S, Crumpacker CS. Prognostic value of plasma human immunodeficiency virus type 1 (HIV-1) RNA levels in patients with advanced HIV-1 disease and with little or no prior zidovudine therapy. AIDS Clinical Trials Group Protocol 116A/116B/117 Team. J Infect Dis. 1996 Oct;174(4):696-703. doi: 10.1093/infdis/174.4.696. PMID 8843205
- [Result] Coombs RW, Welles SL, Hooper C, Reichelderfer PS, D'Aquila RT, Japour AJ, Johnson VA, Kuritzkes DR, Richman DD, Kwok S, Todd J, Jackson JB, DeGruttola V, Crumpacker CS, Kahn J. Association of plasma human immunodeficiency virus type 1 RNA level with risk of clinical progression in patients with advanced infection. AIDS Clinical Trials Group (ACTG) 116B/117 Study Team. ACTG Virology Committee Resistance and HIV-1 RNA Working Groups. J Infect Dis. 1996 Oct;174(4):704-12. doi: 10.1093/infdis/174.4.704. PMID 8843206
- [Result] Mildvan D, Spritzler J, Grossberg SE, Fahey JL, Johnston DM, Schock BR, Kagan J. Serum neopterin, an immune activation marker, independently predicts disease progression in advanced HIV-1 infection. Clin Infect Dis. 2005 Mar 15;40(6):853-8. doi: 10.1086/427877. Epub 2005 Feb 18. PMID 15736019